CLINICAL TRIAL: NCT04667936
Title: Evaluation of Impaired Sedation in Patients With Moderate to Severe COVID-19 ARDS
Brief Title: Evaluation of Sedation in COVID-19 ARDS
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Elisabeth H. Adam, Senior Physician, Goethe University
Other Study IDs: #20-643 -Sed II
Record Dates: First submitted 2020-11-25; First posted 2020-12-16 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Prone Position; Severe Acute Respiratory Syndrome Coronavirus 2; Hypnotics and Sedatives; Pulmonary Ventilation
Keywords: Critical Care; acute respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- moderate to severe COVID-19 ARDS: patients with an oxygenation index <200 under intubation anesthesia and mechanical ventilation.
  Interventions: Other: Treatment group

INTERVENTIONS:
Other: Treatment group — None, solely treatment documentation

SUMMARY:
This study focuses on the evaluation of various factors repeatedly discussed in relation to the impaired sedation of intubated ventilated COVID-19 patients. The sedation response of >100 moderately to severely affected COVID-19 ARDS was evaluated. The sedation level was measured at the bedside using the Richmond Agitation and Sedation Scale and ventilator synchrony. The evaluation was performed according to the static evaluation plan with respect to age, storage therapy and organ failure.

ELIGIBILITY:
Inclusion Criteria:

moderate to severe COVID-19 ARDS

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients admitted to the intensive care unit who were already diagnosed with (SARS-CoV-2) infection.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Position therapy | Data collection is performed at the date of death from any cause or discharge up to 10 weeks.
  Number of positioning therapys during treatment
Agitation and sedation level | 30 minutes after study enrolment
  Measurement is performed using the Richmond Agitation and Sedation Scale (RASS, range: -5[Unarousable] to +4 [Combative], normal condition=0 [Alert and calm])
Agitation and sedation level | Change in average dosage within 8 hours.
  Change of sedation level using the Richmond Agitation and Sedation Scale (RASS, range: -5[Unarousable] to +4 [Combative], normal condition=0 [Alert and calm])
Application of opioid analgesic | 30 minutes after study enrolment
  Applied dosage of sufentanil (measured in µg/kg/h)
Change of application of opioid analgesic | Change in average dosage within 8 hours.
  Applied dosage of sufentanil (measured in µg/kg/h)
Application of opioid analgesic | 30 minutes after study enrolment
  Applied dosage of remifentanil (measured in µg/kg/min)
Change of application of opioid analgesic | Change in average dosage within 8 hours.
  Applied dosage of remifentanil (measured in µg/kg/min)
Application of sedative | 30 minutes after study enrolment
  Applied dosage of midazolam (measured in mg/kg/h)
Change in sedative dosage applied | Change in average dosage within 8 hours.
  Applied dosage of midazolam (measured in mg/kg/h)
Application of sedative | 30 minutes after study enrolment
  Applied dosage of propofol (measured in mg/kg/h)
Change in sedative dosage applied | Change in average dosage within 8 hours.
  Applied dosage of propofol (measured in mg/kg/h)
Application of sedative | 30 minutes after study enrolment
  Applied dosage of lormetazepam (measured in mg/kg/min)
Change in sedative dosage applied | Change in average dosage within 8 hours.
  Applied dosage of lormetazepam (measured in mg/kg/min)
Application of sedative | 30 minutes after study enrolment
  Applied dosage of clonidine (measured in µg/kg/h)
Change in sedative dosage applied | Change in average dosage within 8 hours.
  Applied dosage of clonidine (measured in µg/kg/h)
Application of sedative | 30 minutes after study enrolment
  Applied dosage of Dexmethomidine (measured in µg/kg/h)
Change in sedative dosage applied | Change in average dosage within 8 hours.
  Applied dosage of Dexmethomidine (measured in µg/kg/h)
Application of sedative | 30 minutes after study enrolment
  Applied dosage of esketamine (measured in mg/kg/h)
Change in sedative dosage applied | Change in average dosage within 8 hours.
  Applied dosage of esketamine (measured in mg/kg/h)
Patient Characteristics | The data is recorded at the time of enrolment
  Age (in years)
Patient Characteristics | The data is recorded at the time of enrolment
  Height (in centimeters)
Patient Characteristics | The data is recorded at the time of enrolment
  Weight (in kilograms)

SECONDARY OUTCOMES:
Need for renal replacement therapy | Data collection is performed at the date of death from any cause or discharge up to 10 weeks.
  The necessity and application of a renal replacement procedure is documented
Need for extracorporeal membrane oxygenation (vvECMO) | Data collection is performed at the date of death from any cause or discharge up to 10 weeks.
  The necessity and application of an extracorporeal oxygenation procedure (ECMO) is documented

CONTACTS AND LOCATIONS:
Overall Officials: Armin N Flinspach, MD, Principal Investigator — KGU
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No